CLINICAL TRIAL: NCT02742727
Title: Chimeric Antigen Receptor-Modified pNK Cells for CD7 Positive Relapsed or Refractory Leukemia and Lymphoma
Brief Title: CAR-pNK Cell Immunotherapy in CD7 Positive Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Hefei (Other); Hefei Binhu Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-107-002
Record Dates: First submitted 2016-03-31; First posted 2016-04-19 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acute Myeloid Leukemia; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; T-cell Prolymphocytic Leukemia; T-cell Large Granular Lymphocytic Leukemia; Peripheral T-cell Lymphoma, NOS; Angioimmunoblastic T-cell Lymphoma; Extranodal NK/T-cell Lymphoma, Nasal Type; Enteropathy-type Intestinal T-cell Lymphoma; Hepatosplenic T-cell Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic, T-Cell; Leukemia, Large Granular Lymphocytic; Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Extranodal NK-T-Cell; Enteropathy-Associated T-Cell Lymphoma | interventions — Sensitivity and Specificity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-pNK Cell immunotherapy (Experimental): Enrolled patients will receive CAR-pNK cell immunotherapy with a novel specific chimeric antigen receptor targeting CD7 antigen by infusion.
  Interventions: Biological: anti-CD7 CAR-pNK cells

INTERVENTIONS:
Biological: anti-CD7 CAR-pNK cells — The allogeneic NK cells (NK-92 cell line for clinical use) are engineered to contain anti-CD7 attached to TCRzeta, CD28 and 4-1BB signaling domains. These modified cells are called chimeric antigen receptor NK cells with specificity for CD7.
  Other Names: chimeric antigen receptor NK cells with specificity for CD7

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CAR-pNK cell immunotherapy in patients with CD7 positive relapsed or refractory Leukemia and Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with CD7+ malignancies in patients with no available curative treatment options who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled:

1. Eligible diseases: CD7 positive relapsed or refractory Leukemia and Lymphoma. ￚ Acute myeloid leukemia, previously identified as CD7+ ￚ Precursor T lymphoblast leukemia/lymphoma ￚ T-cell prolymphocytic leukemia ￚ T-cell large granular lymphocytic leukemia ￚ Peripheral T-cell lymphoma, NOS ￚ Angioimmunoblastic T-cell lymphoma ￚ Extranodal NK/T-cell lymphoma, nasal type ￚ Enteropathy-type intestinal T-cell lymphoma ￚ Hepatosplenic T-cell lymphoma
2. Patients 18 years of age or older, and must have a life expectancy > 12 weeks.
3. CD7 is expressed in malignancy tissues by immuno-histochemical (IHC) or Flow cytometry.
4. Assessable disease as measured by laboratory and bone marrow examinations.
5. Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.
6. Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR-pNK cells.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
8. Ability to give informed consent.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) involvement.
2. Pregnant or nursing women may not participate.
3. Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
5. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
6. Previously treatment with any gene therapy products.
7. The existence of unstable or active ulcers or gastrointestinal bleeding.
8. Patients with a history of organ transplantation or are waiting for organ transplantation.
9. Patients need anticoagulant therapy (such as warfarin or heparin).
10. Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-CD7 CAR-pNK cells | 2 years
  Determine the toxicity profile of the CD7 targeted CAR-pNK cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Clinical response to CD7 CAR-pNK cell infusions | Safety follow-up is 100 days from last CAR-pNK infusion
  Patients with measurable disease will be assessed for the response of their disease to CD7 CAR-pNK cell treatment.
Determine the existence of CD7-CAR-pNK in vivo | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Ph.D., Principal Investigator — PersonGen BioTherapeutics (Suzhou) Co., Ltd.
Locations (1):
- PersonGen BioTherapeutics (Suzhou) Co., Ltd., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Del Zotto G, Marcenaro E, Vacca P, Sivori S, Pende D, Della Chiesa M, Moretta F, Ingegnere T, Mingari MC, Moretta A, Moretta L. Markers and function of human NK cells in normal and pathological conditions. Cytometry B Clin Cytom. 2017 Mar;92(2):100-114. doi: 10.1002/cyto.b.21508. Epub 2017 Feb 12. PMID 28054442